CLINICAL TRIAL: NCT01919528
Title: Real-time Ultrasound-guided Catheterization of the Axillary Vein in the Intensive Care Unit
Brief Title: Ultrasound-guided Catheterization of the Axillary Vein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Tomasz Czarnik, MD PhD, senior anesthesiologist, Uniwersytecki Szpital Kliniczny w Opolu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Axillary-US-guided-1; Axillary-1 (Other: PS ZOZ Wojewodzkie Centrum Medyczne w Opolu)
Record Dates: First submitted 2013-08-04; First posted 2013-08-09 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Critical Illness
Keywords: ultrasonography; catheterization; central line; mechanical ventilation; intensive care; axillary vein
MeSH Terms: conditions — Critical Illness | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- axillary vein catheterization (Experimental): central venous catheter placement into the axillary vein under ultrasound guidance
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — catheterization of the axillary vein under ultrasound guidance

SUMMARY:
The central venous catheterization (central line placement) is the common procedure performed in the intensive care unit. This procedure is performed by percutaneous puncture of so called 'the central vein' and than advancement of the catheter over the guidewire (Seldinger technique). The tip of the catheter is left in the superior vena cava in the vicinity of the right atrium of the heart. Central veins are large veins in the human body passing the blood into the heart.

Typical, clinical indications for the central line placement in the intensive care unit are hemodynamic monitoring, volume monitoring, administration of medications, long-term total parenteral nutrition, access for renal replacement therapy, difficult peripheral catheterization.

There are two methods of the central venous catheterization in terms of visualization. First and older is the blind technique. The operator is locating the anatomical landmarks and then performing the entire procedure blindly by percutaneous puncture. This is called the landmark technique. Second and new is the ultrasound-guided technique. The operator is locating the vein using ultrasonography and then performing the entire procedure under ultrasonographic visualization. The real time ultrasound-guided central venous catheterization became the standard of care in recent years mainly because of safety issues (is regarded as safer than landmark technique)

The catheterization of the axillary vein is not popular procedure in daily clinical practice. But it can be reasonable and safe alternative to others, typically performed central venous catheterizations like the internal jugular vein and the subclavian vein catheterizations.

The main intention of this study is to assess usefulness and safety of the real time ultrasound guided axillary vein catheterization in mechanically ventilated patients admitted to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated intensive care patients with clinical indications for central venous line placement

Exclusion Criteria:

* trauma and hematoma at the catheterization site
* history of multiple central venous catheterizations (three or more)
* chest wall deformities
* major blood coagulation disorders
* history of thoracic surgery
* anatomical abnormalities at the catheterization site
* infection at the catheterization site
* age less than 18 years
* lack of patients or closest relatives consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
to define venipuncture, catheterization and entire procedure success rates | 24 hours
  the venipuncture is defined as perforation of the axillary vein by the needle, the catheterization is defined as the placement of catheter in the final position, the entire procedure success rate is defined as the placement of catheter in the final position without early complications (assessed within 24 hours time frame)
to assess the erly complication rate of ultrasound-guided axillary vein catheterization | 24 hours
  pneumothorax, puncture of the axillary artery, hemothorax, heart perforation, catheter malposition, significant arrhythmias, air embolism

SECONDARY OUTCOMES:
to assess the correlation between entire procedure success rate and the side of catheterization | 2 years
  the left axillary vein or the right axillary vein
to assess the correlation between patients weight, height and depth, diameter of the axillary vein | 2 years
  the depth and diameter of the axillary vein is measured by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Czarnik, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, Publiczny Samodzielny Zaklad Opieki Zdrowotnej Wojewodzkie Centrum Medyczne w Opolu
Locations (1):
- Department of Anesthesiology and Intensive Care, Publiczny Samodzielny Zaklad Opieki Zdrowotnej Wojewodzkie Centrum Medyczne w Opolu, Opole, Poland

REFERENCES:
- [Result] Czarnik T, Gawda R, Nowotarski J. Real-time, ultrasound-guided infraclavicular axillary vein cannulation for renal replacement therapy in the critical care unit-A prospective intervention study. J Crit Care. 2015 Jun;30(3):624-8. doi: 10.1016/j.jcrc.2015.01.002. Epub 2015 Jan 8. PMID 25697988
- [Result] Czarnik T, Gawda R, Nowotarski J. Real-time ultrasound-guided infraclavicular axillary vein cannulation: A prospective study in mechanically ventilated critically ill patients. J Crit Care. 2016 Jun;33:32-7. doi: 10.1016/j.jcrc.2016.02.021. Epub 2016 Mar 2. PMID 26993368